CLINICAL TRIAL: NCT01315756
Title: The Norwegian Study in Renewing Health: Stimulating Self-management in Patients With Type 2 Diabetes Mellitus Through Telecare With the Few Touch Application and Health Counseling - a Randomized Controlled Trial
Brief Title: Self-management in Type 2 Diabetes Patients Using the Few Touch Application
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: Oslo University College (Other); European Commission (Other); The Research Council of Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Renewing Health Norway
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (No Intervention): Treatment as usual.
- Few Touch Application (FTA) (Experimental): This arm will receive a Smartphone with the diabetes diary application ("the Few Touch application"), a self-help tool that consists of five main elements accessible to the user.
  Interventions: Device: Use of Few Touch Application (FTA)
- FTA and health counseling (Experimental): This arm will additionally receive health counseling based on TTM and CBT by a diabetes nurse with individualized feedback via sms from the diabetes nurse which is based on the patient's initiative (via sms). In addition, the diabetes nurse will call the patients three times during this period and discuss progress.
  Interventions: Device: Use of FTA and health counseling based on TTM and CBT

INTERVENTIONS:
Device: Use of Few Touch Application (FTA) — The users will receive a Smartphone with the diabetes diary application ("the Few Touch application"), a self-help tool that consists of five main elements accessible to the user. The five elements are the food habits registration, blood glucose data management system, physical activity registration, personal goals setting and general information. While blood glucose data is automatically transferred to the phone from the blood glucose meter when the user has performed a measurement, activity data and food habits have to be entered manually by the user.
  Other Names: Use of Diabetesdagbok
  Arms: Few Touch Application (FTA)
Device: Use of FTA and health counseling based on TTM and CBT — The users will additionally receive health counseling based on TTM and CBT by a diabetes nurse with individualized feedback via SMS from the diabetes nurse which is based on the patient's initiative (via SMS). In addition, the diabetes nurse will call the patients three times during this period and discuss progress. Both the SMS-messages and the calls will be based on CBT according to the TTM-level. The intervention allows information to be given both in an individualized and tailored manner for each particular patient by the nurse, but also in a general way via SMS. The patients need to understand the relationship between areas such as glucose levels, diet, exercises and medicine, in the context of their own lifestyle needs.
  Other Names: Use of Few Touch Application with Health Counseling
  Arms: FTA and health counseling

SUMMARY:
It is hypothesized that the use of the mobile phone-based self-help system FTA, and with the patients as active players, will improve diabetes self-management reflected by improved glycemic control and lipids, self-care behaviours and lifestyle changes such as improved dietary habits and increased physical activity, compared with usual care. Following this; it is also hypothesized that this will also lead to a reduction in overall risk for diabetes complications (expressed by reduction in e.g., 5 year absolute risk for coronary artery disease as calculated using the Swedish National Diabetes Register's risk calculator) and in the prevalence of the metabolic syndrome (e.g., as defined by the International Diabetes Federation). It also hypothesized that health counselling based on TTM and CBT by a diabetes nurse, and with individualized feedback via sms from the diabetes nurse, may have an important function as a supplement to the self-help system (FTA). In addition, it is hypothesized that the patients' health status and diabetes-related quality of life (HRQL) will improve. The results of this study may show that a commonly used tool like the mobile phone, and also mobile phone together with health counselling, fitted into the patients' daily life, is more effective and cost-effective than standard care.

DETAILED DESCRIPTION:
The purpose of this study is to examine the effectiveness of mobile phone-based lifestyle tools, and health counseling using tailored SMS and individual phone-calls to the patients, for self-management of T2DM. Maintaining daily symptom diaries (described below) by an easy way of self-monitoring appear to offer a valid and reliable way of assessing behaviours. In addition, the patients are able to view their own registrations on the Smartphone, i.e. a programmable mobile phone with a touch sensitive screen. The self-help system, called the "Few Touch application", recently tested on 12 people with T2DM at NST, University Hospital of North Norway (UNN), will form the basis for the patients' mobile interaction system.

ELIGIBILITY:
Inclusion Criteria:

Age >18; diagnosed T2DM > 3 months prior to study inclusion; in case the patient is receiving one or more glucose lowering drug (e.g., metformin, sulphonylurea, glinide, α-glucosidase inhibitor, DPP-IV inhibitor, GLP-1 analogue, glitazone, insulin) the treatment should be stabilized (i.e., no change in dosage the last three months prior to inclusion except for insulin treated patients who are allowed ±15% dose adjustment; HbA1c >7%; capability of understanding and filling in Norwegian questionnaires; be able to use the system provided; be cognitive able to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2011-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Improved glycemic control, HbA1c | One year
  It is hypothesized that the use of the mobile phone-based self-help system FTA, and with the patients as active players, will improve diabetes self-management reflected by improved glycemic control.

SECONDARY OUTCOMES:
Lipids, self-care, lifestyle changes, complications, quality of life. | One year
  It is hypothesized that the use of the mobile phone-based self-help system FTA will improve diabetes self-management, reflected by improved lipids values, self-care behaviors and lifestyle changes compared with usual care, that this will also lead to a reduction in overall risk for diabetes complications, that health counseling based on TTM and CBT by a diabetes nurse and with individualized feedback via SMS may have an important function as a supplement to the self-help system, and that the patients' health status and diabetes-related quality of life will improve.

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Engum, M.Sc. / M.HA, Study Chair — Norwegian Centre for Integrated Care and Telemedicine (NST ), University Hospital of North- Norway
Locations (2):
- Norway (2):
  - Oslo University College, Oslo, Oslo County
  - Norwegian Centre for Integrated Care and Telemedicine (NST ), University Hospital of North- Norway, Tromsø, Troms

REFERENCES:
- [Background] Arsand E, Tatara N, Ostengen G, Hartvigsen G. Mobile phone-based self-management tools for type 2 diabetes: the few touch application. J Diabetes Sci Technol. 2010 Mar 1;4(2):328-36. doi: 10.1177/193229681000400213. PMID 20307393
- [Background] Arsand E, Tufano JT, Ralston JD, Hjortdahl P. Designing mobile dietary management support technologies for people with diabetes. J Telemed Telecare. 2008;14(7):329-32. doi: 10.1258/jtt.2008.007001. PMID 18852310
- [Background] Arsand E, Demiris G. User-centered methods for designing patient-centric self-help tools. Inform Health Soc Care. 2008 Sep;33(3):158-69. doi: 10.1080/17538150802457562. PMID 18850399
- [Background] Wangberg SC, Arsand E, Andersson N. Diabetes education via mobile text messaging. J Telemed Telecare. 2006;12 Suppl 1:55-6. doi: 10.1258/135763306777978515. PMID 16884582
- [Background] Gammon D, Arsand E, Walseth OA, Andersson N, Jenssen M, Taylor T. Parent-child interaction using a mobile and wireless system for blood glucose monitoring. J Med Internet Res. 2005 Nov 21;7(5):e57. doi: 10.2196/jmir.7.5.e57. PMID 16403721
- [Derived] Torbjornsen A, Ribu L, Ronnevig M, Grottland A, Helseth S. Users' acceptability of a mobile application for persons with type 2 diabetes: a qualitative study. BMC Health Serv Res. 2019 Sep 6;19(1):641. doi: 10.1186/s12913-019-4486-2. PMID 31492176
- [Derived] Torbjornsen A, Smastuen MC, Jenum AK, Arsand E, Ribu L. Acceptability of an mHealth App Intervention for Persons With Type 2 Diabetes and its Associations With Initial Self-Management: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2018 May 21;6(5):e125. doi: 10.2196/mhealth.8824. PMID 29784635
- [Derived] Holmen H, Wahl A, Torbjornsen A, Jenum AK, Smastuen MC, Ribu L. Stages of change for physical activity and dietary habits in persons with type 2 diabetes included in a mobile health intervention: the Norwegian study in RENEWING HEALTH. BMJ Open Diabetes Res Care. 2016 May 12;4(1):e000193. doi: 10.1136/bmjdrc-2016-000193. eCollection 2016. PMID 27239317
- [Derived] Ribu L, Holmen H, Torbjornsen A, Wahl AK, Grottland A, Smastuen MC, Elind E, Bergmo TS, Breivik E, Arsand E. Low-intensity self-management intervention for persons with type 2 diabetes using a mobile phone-based diabetes diary, with and without health counseling and motivational interviewing: protocol for a randomized controlled trial. JMIR Res Protoc. 2013 Aug 26;2(2):e34. doi: 10.2196/resprot.2768. PMID 23978690